CLINICAL TRIAL: NCT06160700
Title: Serial Testing To Assess Cognitive Function In Patients With Cancer Being Treated With Immunotherapy
Brief Title: Serial Testing To Assess Cognitive Function In Cancer
Status: Terminated | Type: Observational
Why Stopped: loss of research support
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Nasser Hanna, Professor of Medicine, Associate Division Director of Oncology, Indiana University
Other Study IDs: CTO-IUSCCC-0770
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Cancer
Keywords: Cancer; Immunotherapy; Cognitive Assessment; Montreal Cognitive Assessment; Chemo Brain
MeSH Terms: conditions — Neoplasms | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Immunotherapy Only: Subjects who are currently receiving immunotherapy only.
  Interventions: Behavioral: Montreal Cognitive Assessment (MoCA)
- Chemo-Immunotherapy Control Arm: Subjects who are receiving chemo-immunotherapy.
  Interventions: Behavioral: Montreal Cognitive Assessment (MoCA)
- No Active Therapy Control Arm: Subjects who are no currently receiving active therapy.
  Interventions: Behavioral: Montreal Cognitive Assessment (MoCA)

INTERVENTIONS:
Behavioral: Montreal Cognitive Assessment (MoCA) — MoCA is a method for evaluating cognition. This assessment will be conducted at baseline, month 3, and month 6.

SUMMARY:
The purpose of this study is to examine the effects of immunotherapy on cognitive function of cancer patients and follow them clinically over a period of six months with the Montreal cognitive assessment (MoCA) to assess changes in cognition.

DETAILED DESCRIPTION:
"Chemo brain" has been described as a side effect of conventional chemotherapy and radiotherapy in cancer patients. With the advent of immunotherapy and progress made in treatment of cancer, long term-survival has increased which raises the question of preserving cognitive function in these patients. However, to date, no large center studies have been done to assess the effects of immunotherapy on cognitive function in patients of all cancer types. Studies that have been done are on preclinical models and very small number of patients, which remained inconclusive.

The primary objective of this pilot clinical trial is to estimate the rate of cognitive function change using the MoCA scale over 6 months in each individual group of patients with cancer treated with immunotherapy alone, combined chemotherapy and immunotherapy, and in patients with cancer on no active treatment, respectively. The secondary objective is to estimate the changes of MoCA scores after 3 months and 6 months in patients receiving immunotherapy alone for the treatment of their cancer.

ELIGIBILITY:
Inclusion Criteria for Immunotherapy Only Group:

1. Age ≥ 18 years old
2. Ability to provide written informed consent and HIPAA authorization.
3. Patients with any type or stage of cancer eligible to begin treatment with immunotherapy alone.

Note: Prior radiation therapy if not to the brain is acceptable.

Inclusion Criteria for Chemotherapy plus Immunotherapy Control Arm:

1. Age ≥ 18 years old
2. Ability to provide written informed consent and HIPAA authorization.
3. Patients with any stage of cancer eligible to begin treatment with chemoimmunotherapy.

Note: Prior radiation therapy if not to the brain is acceptable.

Note: Patients receiving chemotherapy followed by immunotherapy between baseline and the 3 months MoCA will be eligible.

Inclusion Criteria for Patients not on Active Treatment Control Arm:

1. Age ≥ 18 years old
2. Ability to provide written informed consent and HIPAA authorization.
3. Patients with a prior history of cancer treated with surgery alone at least 1 year out of treatment OR surgery and neo-adjuvant/adjuvant chemotherapy who are at least 2 years out from treatment. If patients underwent any other form of treatment for their current malignancy, they will be excluded.

Note: Prior radiation therapy if not to the brain is acceptable.

Exclusion Criteria:

1. Patients who screen positive for depression by PHQ-2 test defined as a score more than 3 will complete the PHQ-9 questionnaire. If they screen positive for depression on the PHQ-9 questionnaire (score of 10 or more) or refuse to complete it, they will be excluded.
2. Patients with a history of prior malignancy (excluding skin squamous cell or basal cell cancers).
3. Patients with history of brain radiation and brain metastasis.
4. Patients with a known prior diagnosis of cognitive dysfunction such as dementia from either Alzheimer's, vascular dementia, Parkinson's, mental retardation, head injury etc. Or any uncontrolled etiologies that can affect cognitive function such as anxiety, depression, bipolar disorder, schizophrenia and hypo/hyperthyroidism will be excluded.

Note: patients with controlled anxiety/ depression who don't screen positive on the PHQ-2 scale are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a prospective single site pilot study enrolling subjects with any stage of cancer who are receiving immunotherapy as part of their treatment. Subjects will be recruited from the clinics of the IUSCCC and Eskenazi Health. Subjects will be matched into three groups based on demographics including age, sex and self-reported educational level.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Rate of Cognitive Function Change | Baseline and 6 months
  The changes in MoCA scores over 6 months in patients from each group will be plotted and summarized with mean change, standard deviation of change, and standard errors of mean change. The standardized response mean (SRM), calculated as the mean change from baseline to 6 months, divided by the standard deviation of change, will be reported as the main effect size for evaluating the magnitude of change in cognitive function.

SECONDARY OUTCOMES:
Changes in MoCA scores | 3 and 6 months
  Changes of MoCA scores at 3 months and 6 months from the immunotherapy group will be fitted by the mixed-effects linear model including time effects, which will describe the relationship between the common effect of MoCA score changes, the random effect of time, and the random error representing subjects' observation time.

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Hanna, MD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana